CLINICAL TRIAL: NCT02644655
Title: A Clinical Study Using Autologous T Cell Engineered With Chimeric Antigen Receptor Targeting to CD19（Cluster of Differentiation Antigen 19) in Treating Patients With Recurrent /Refractory B Cell Leukemia
Brief Title: Immunotherapy Using Autologous T Cell-Engineered With CD19-specific Chimeric Antigen Receptor for the Treatment of Recurrent /Refractory B Cell Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2015-02-007
Record Dates: First submitted 2015-12-12; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-09

CONDITIONS: Recurrent B-Cell Tumor; Refractory B-Cell Tumor
Keywords: Recurrent B-Cell Tumor; Refractory B-Cell Tumor; New Cluster of Differentiation Antigen 19-chimeric Antigen Receptor T Cells; safety; prognosis
MeSH Terms: interventions — CD19-specific chimeric antigen receptor

ARMS (1):
- CD19-specific chimeric antigen receptor (Experimental): After pretreatment, cluster of differentiation antigen 19 (CD19)-specific chimeric antigen receptor will be transfused.
  Interventions: Biological: CD19-specific chimeric antigen receptor

INTERVENTIONS:
Biological: CD19-specific chimeric antigen receptor — Cyclophosphamide 500 mg - 2000 mg/m2 (day 2) with or without Fludarabine 30 mg/m2 /day, 4 days (day 6, 5, 4, 3); nCAR19-T transfusion：day 0(5×105/kg，1×106/kg，3×106/kg).

SUMMARY:
Objectives:

The purpose of this study is to evaluate the safety and prognosis of New Cluster of Differentiation Antigen 19-chimeric Antigen Receptor T (nCAR19-T) Cells in the treatment of recurrent/refractory B-cell tumor and the Optimal dosage of nCAR19-T cell therapy.

Methods:

This study designs a novel therapy using nCAR19-T. 20 patients will be enrolled. Cyclophosphamide 500 mg - 2000 mg/m2 (day 2) with or without Fludarabine 30 mg/m2 /day, 4 days (day-6,-5,-4,-3); nCAR19-T transfusion：day 0(5×10※5/kg，1×10※6/kg，3×10※6/kg). According to the National Cancer Institute (NCI) standard (CTCAE), they will be observed 24 weeks long. Follow-up survey after the clinical study: within 1 months, once a week; then once a month for 1 years; and then once a year, a total of 15 years.

DETAILED DESCRIPTION:
A total of 20 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female
2. Karnofsky≥60%
3. At least 2 courses of chemotherapy were performed
4. Creatinine is less than 2.5mg/dL;alanine aminotransferase (ALT) / aspartate aminotransferase(AST) less than 3 times of the normal bilirubin is less than 3mg/dL
5. Adequate venous access, isolation, and white blood cell production without other taboos
6. Signed informed consent
7. Patients with fertility are willing to use contraceptive method.
8. At least two months after infusion of T cells

Exclusion Criteria:

1. Need to use glucocorticoid therapy
2. Need immunotherapy
3. Creatinine > 2.5mg/dL; ALT / AST > 5 times of the normal; bilirubin > 3mg/dL
4. Forced expiratory volume at one second (FEV1)<2 L,diffusing capacity of the lung for carbon monoxide (DLCO)<40%
5. congestive cardiac failure (III or IV, NYHA); Significant hypotension; Coronary heart disease Can not be controlled; DLCO<40%
6. human immunodeficiency virus (HIV), hepatitis B virus (HBV),hepatitis C virus (HCV) patients
7. Had received gene therapy
8. Significant encephalopathy / new focal neurologic impairment
9. Blood culture positive or radiographic evidence of infection
10. Other drugs, or other biological treatment, chemotherapy or radiotherapy are performed within a month
11. The history of allergic reactions in cell therapy and cetuximab similar compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events and tumor response rate related to study drug | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Qian, PHD, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China

REFERENCES:
- [Background] Ghorashian S, Pule M, Amrolia P. CD19 chimeric antigen receptor T cell therapy for haematological malignancies. Br J Haematol. 2015 May;169(4):463-78. doi: 10.1111/bjh.13340. Epub 2015 Mar 5. PMID 25753571
- [Background] Maude SL, Shpall EJ, Grupp SA. Chimeric antigen receptor T-cell therapy for ALL. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):559-64. doi: 10.1182/asheducation-2014.1.559. Epub 2014 Nov 18. PMID 25696911
- [Background] Grupp SA. Advances in T-cell therapy for ALL. Best Pract Res Clin Haematol. 2014 Sep-Dec;27(3-4):222-8. doi: 10.1016/j.beha.2014.10.014. Epub 2014 Oct 27. PMID 25455270
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Background] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870
- [Background] Kochenderfer JN, Dudley ME, Kassim SH, Somerville RP, Carpenter RO, Stetler-Stevenson M, Yang JC, Phan GQ, Hughes MS, Sherry RM, Raffeld M, Feldman S, Lu L, Li YF, Ngo LT, Goy A, Feldman T, Spaner DE, Wang ML, Chen CC, Kranick SM, Nath A, Nathan DA, Morton KE, Toomey MA, Rosenberg SA. Chemotherapy-refractory diffuse large B-cell lymphoma and indolent B-cell malignancies can be effectively treated with autologous T cells expressing an anti-CD19 chimeric antigen receptor. J Clin Oncol. 2015 Feb 20;33(6):540-9. doi: 10.1200/JCO.2014.56.2025. Epub 2014 Aug 25. PMID 25154820
- [Background] Davila ML, Riviere I, Wang X, Bartido S, Park J, Curran K, Chung SS, Stefanski J, Borquez-Ojeda O, Olszewska M, Qu J, Wasielewska T, He Q, Fink M, Shinglot H, Youssif M, Satter M, Wang Y, Hosey J, Quintanilla H, Halton E, Bernal Y, Bouhassira DC, Arcila ME, Gonen M, Roboz GJ, Maslak P, Douer D, Frattini MG, Giralt S, Sadelain M, Brentjens R. Efficacy and toxicity management of 19-28z CAR T cell therapy in B cell acute lymphoblastic leukemia. Sci Transl Med. 2014 Feb 19;6(224):224ra25. doi: 10.1126/scitranslmed.3008226. PMID 24553386
- [Background] Maher J. Clinical immunotherapy of B-cell malignancy using CD19-targeted CAR T-cells. Curr Gene Ther. 2014 Feb;14(1):35-43. doi: 10.2174/1566523213666131223130554. PMID 24365143
- [Background] Cheadle EJ, Gornall H, Baldan V, Hanson V, Hawkins RE, Gilham DE. CAR T cells: driving the road from the laboratory to the clinic. Immunol Rev. 2014 Jan;257(1):91-106. doi: 10.1111/imr.12126. PMID 24329792
- [Background] Kochenderfer JN, Dudley ME, Carpenter RO, Kassim SH, Rose JJ, Telford WG, Hakim FT, Halverson DC, Fowler DH, Hardy NM, Mato AR, Hickstein DD, Gea-Banacloche JC, Pavletic SZ, Sportes C, Maric I, Feldman SA, Hansen BG, Wilder JS, Blacklock-Schuver B, Jena B, Bishop MR, Gress RE, Rosenberg SA. Donor-derived CD19-targeted T cells cause regression of malignancy persisting after allogeneic hematopoietic stem cell transplantation. Blood. 2013 Dec 12;122(25):4129-39. doi: 10.1182/blood-2013-08-519413. Epub 2013 Sep 20. PMID 24055823
- [Background] Grupp SA, Kalos M, Barrett D, Aplenc R, Porter DL, Rheingold SR, Teachey DT, Chew A, Hauck B, Wright JF, Milone MC, Levine BL, June CH. Chimeric antigen receptor-modified T cells for acute lymphoid leukemia. N Engl J Med. 2013 Apr 18;368(16):1509-1518. doi: 10.1056/NEJMoa1215134. Epub 2013 Mar 25. PMID 23527958
- [Background] Brentjens RJ, Davila ML, Riviere I, Park J, Wang X, Cowell LG, Bartido S, Stefanski J, Taylor C, Olszewska M, Borquez-Ojeda O, Qu J, Wasielewska T, He Q, Bernal Y, Rijo IV, Hedvat C, Kobos R, Curran K, Steinherz P, Jurcic J, Rosenblat T, Maslak P, Frattini M, Sadelain M. CD19-targeted T cells rapidly induce molecular remissions in adults with chemotherapy-refractory acute lymphoblastic leukemia. Sci Transl Med. 2013 Mar 20;5(177):177ra38. doi: 10.1126/scitranslmed.3005930. PMID 23515080
- [Background] Terakura S, Yamamoto TN, Gardner RA, Turtle CJ, Jensen MC, Riddell SR. Generation of CD19-chimeric antigen receptor modified CD8+ T cells derived from virus-specific central memory T cells. Blood. 2012 Jan 5;119(1):72-82. doi: 10.1182/blood-2011-07-366419. Epub 2011 Oct 26. PMID 22031866
- [Background] Porter DL, Levine BL, Kalos M, Bagg A, June CH. Chimeric antigen receptor-modified T cells in chronic lymphoid leukemia. N Engl J Med. 2011 Aug 25;365(8):725-33. doi: 10.1056/NEJMoa1103849. Epub 2011 Aug 10. PMID 21830940